CLINICAL TRIAL: NCT05621746
Title: Non-Interventional Study of the Change in Joint Health in Adult Patients With Haemophilia A After Switching to Prophylaxis With Turoctocog Alfa Pegol (N8-GP)
Brief Title: An Observational Research Study of the Health of Joints in People With Haemophilia Taking the Medicine Esperoct
Status: Recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7088-4928; U1111-1271-9209 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Haemophilia A: Participants will be treated with commercially available Esperoct for a total study duration of 24 months according to the local label and local routine clinical practice at the discretion of the physician. The decision to switch to Esperoct will be made prior to and separate from the decision to enrol in the study.
  Interventions: Drug: Esperoct

INTERVENTIONS:
Drug: Esperoct — Participants will be treated with commercially available Esperoct for a total study duration of 24 months according to the local label and local routine clinical practice at the discretion of the physician. The decision to switch to Esperoct will be made prior to and separate from the decision to enrol in the study.
  Other Names: Turoctocog alfa pegol (N8-GP)

SUMMARY:
This study will collect information on the long term health of joints in people with haemophilia A who have started treatment with Esperoct within twelve months prior to participation to the study. This study is conducted to look at how joint health of people with haemophilia changes over time when they are receiving the medicine Esperoct. The participants will get Esperoct as prescribed to the participants by the study doctor. The participant's treatment will not be affected by their involvement in the study. Every six months, the participants will be asked to answer some questionnaires about their joints, their pain and their ability to be physically active. Their participation in the study will last for no more than 2 years. The participants are free to leave the study at any time and for any reason. This will not affect their current and future medical care.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male, greater than or equal to 18 years of age at the time of signing informed consent, diagnosed with severe (FVIII activity below 1%) or moderate congenital haemophilia A (FVIII activity 1-5%).
* The decision to initiate treatment with commercially available Esperoct has been made by the patient and the treating physician before and independently from the decision to include the patient in this study.
* Switched, within two months prior to enrolment, OR planned to switch, within one month post enrolment, to prophylaxis treatment with Esperoct from previous therapy; the decision to initiate treatment with Esperoct must be made prior to and independently from the decision to enrol in the study.
* Must have baseline data (HJHS, target joints, and medical history) collected in routine clinical practice within two months prior or up to one month post switch to Esperoct therapy.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Previous terminated treatment regimen with Esperoct prophylaxis.
* Current or previously terminated treatment regimen with Esperoct on-demand.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Previous participation in a clinical trial within the 30 days prior to switching to Esperoct.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Participants with Haemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in haemophilia joint health score (HJHS) | From date of switch to end of study (up to 24 months)
  Measured as units on a score. The scoring range of the HJHS is from 0 (normal, healthy joints) to 124 (maximum severity). A sustained HJHS is defined as a change in total score of less than or equal to (<=) 2 points over 24 months.

SECONDARY OUTCOMES:
The number of bleeding episodes requiring coagulation Factor VIII (FVIII) treatment | From baseline to end of study (up to 24 months)
  Measured as episodes
Number of target joints | From baseline to end of study (up to 24 months)
  Measured as number of target joints. Target joints is defined according to the International Society on Thrombosis and Haemostasis (ISTH) as any joint with greater than or equal to (>=) 3 bleeding episodes in the same joint within a 6-month period.
Resolution of any target joints (Yes/No) | From baseline to end of study (up to 24 months)
  Measured as number of resolutions. Target joint resolution is defined according to the ISTH as previously diagnosed target joint that has <=2 spontaneous bleeds in the target joint over 12 month.
Change in patient reported Problem Joint score | From baseline to end of study (up to 24 months)
  Measured in score of problem joints (PJs). A PJ is defined as having chronic joint pain and/or limited range of movement due to compromised joint integrity (i.e. chronic synovitis and/or hemophilic arthropathy). PJ scores are stratified: none, 1 PJ, and 2+ PJs.
Change in patient reported pain scores (Brief Pain Inventory) | From baseline to end of study (up to 24 months)
  Measured as units on a score. The BPI assesses pain at its "worst," "least," "average," and "current pain".
Change in physical function and activity measured using patient reported outcome questionnaires (Short Form-36) | From baseline to end of study (up to 24 months)
  Measured as units on a score. Short form-36 (SF-36) is a 36-item patient-reported survey of patient health that measures the participants's overall health-related quality of life (HRQoL). Scores range from 0-100 (where higher scores indicate a better HRQoL)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency' dept. 2834, Study Director — Novo Nordisk A/S'
Locations (1):
- Novo Nordisk Investigational Site, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com